CLINICAL TRIAL: NCT02143921
Title: Impact of an NGO Training and Support Intervention on Private Sector Provider Diarrhea Management Practices
Brief Title: Impact of Training on Diarrhoea Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2007-051
Record Dates: First submitted 2014-05-18; First posted 2014-05-21 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Acute Childhood Diarrhea
Keywords: NGO zinc scale; compliance with WHO zinc treatment recommendations

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training Intervention (Experimental): One service provider group received training
  Interventions: Behavioral: Training intervention
- Control (No Intervention): Control group service providers did not received intervention training

INTERVENTIONS:
Behavioral: Training intervention — Intervention group service providers received intervention training
  Arms: Training Intervention

SUMMARY:
Alternative, sustainable interventions in support of zinc treatment for childhood diarrhea need to be identified. Within the NGO sector, direct provision of health services is provided, however some NGOs also work closely with the private sector providers. Hypothetically, this avoids unnecessary duplication of effort and enhances the quality of the care provided in the private sector. This study will provide objective evidence of the impact of this approach, using the scale-up of zinc for the treatment of childhood diarrhoea as a test case. The study will be assessing NGO impact among unregulated (unlicensed), rural service providers. Further, this study will serve to assess the value of this model of scaling up activities in the non-state sector with a particular eye toward more generalizable and replicable improvement in quality of care strategies between NGOs and unlicensed private providers. This will be controlled before-after (CBA) study. An equivalent control area will be included in the study. The objective is to document changes in zinc and antibiotic as well as anti-diarrhoeal usage in childhood diarrhea following a scale-up intervention package delivered by a local NGO to local private providers. This will include sensitization, training and follow-up support. Impact will be assessed in terms of changes in zinc coverage and antibiotic use among households in the catchment population served by these providers. The study will be conducted in four unions located in Sreepur Upazila within Gazipur district, located north to Dhaka. Two of the unions, namely Rajabari and Prohladpur comprising 55 villages with 15,530 households and an estimated 76,150 population will serve as intervention area. The other two unions Telihat and Barmi will be taken as control sites. They contain 53 villages with 19,898 households and an estimated 99,000 population. The curative health services in these sites are provided by local drug vendors, village practitioners, traditional healers, and licensed government, private or NGO health service providers. Data will be collected through survey and in-depth interviews. Data will be entered and analyzed using SPSS version 12.0. Absolute counts, proportions, and means with 95% confidence interval will be calculated. These and regression analysis will be done using STATA version 9, cluster survey program, that accounts for potential within cluster homogeneity. Based upon the household surveys, the outcomes that will be calculated are: coverage-the proportion receiving zinc, ORS (zinc and ORS), and antibiotics or antidiarrhoeals and changes in coverage 6 months following the introduction of the intervention package, equity: who is receiving zinc by age, gender and socioeconomic status. For differences in categorical outcomes crude relative risks and 95% confidence intervals will be determined. It is expected that the study will help in increasing zinc coverage for the treatment of children under five years of age and decrease in the use of antibiotics and antidiarrhoeals within the NGO catchment population.

ELIGIBILITY:
Inclusion Criteria:

1. Care takers of the children aged 6 months to 5 years with a prevalent case of diarrhea at the time of the household surveys (within the past 2 weeks). Within each site a systematic household survey will be completed for the identification of any child 6 months to 5 years who has a prevalent case of at least 2 days duration.
2. Health Care Providers

   1. NGO licensed "sub-assistant community medical officers (SACMOs)
   2. Private sector, unlicensed providers: village practitioners and traditional healers

Exclusion Criteria:

N/A

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1160 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To document changes in zinc coverage for acute childhood diarrhoea | 6 months

SECONDARY OUTCOMES:
To document changes in inappropriate use of antibiotics and antidiarrheals | 6 months

OTHER OUTCOMES:
To identify barriers/disincentives to the prescribing of zinc treatment among private providers | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

REFERENCES:
- [Derived] Rahman AS, Islam MR, Koehlmoos TP, Raihan MJ, Hasan MM, Ahmed T, Larson CP. Impact of NGO training and support intervention on diarrhoea management practices in a rural community of Bangladesh: an uncontrolled, single-arm trial. PLoS One. 2014 Nov 14;9(11):e112308. doi: 10.1371/journal.pone.0112308. eCollection 2014. PMID 25398082